CLINICAL TRIAL: NCT00882089
Title: Registry Study of the Contura™ Multi-Lumen Balloon (MLB) Applicator for Accelerated Partial Breast Irradiation in Intermediate-Risk, Pathological Stage 0, I, or II (Up to 3.0 cm) Breast Cancer Patients
Brief Title: Use of the Contura™ Catheter in Intermediate-Risk, Pathological Stage 0, I, or II (Up to 3.0 cm) Breast Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cancer Center of Irvine (Other)
Collaborators: SenoRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1098987
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: Contura; Cancer; Accelerated; Partial; Breast; Irradiation
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): A Contura balloon catheter is placed in the lumpectomy cavity. Later that morning, accelerated partial irradiation begins.
  Interventions: Device: Contura catheter

INTERVENTIONS:
Device: Contura catheter — Radiation therapy is delivered to a total dose of 34 Gy in 10 fractions bid over 5-7 days. Each day, the high dose rate iridium-192 brachytherapy treatments are separated by 6 hours. Each radiation treatment takes 15-30 minutes.
  Other Names: Contura Multi-Lumen Balloon Applicator

SUMMARY:
The purpose of this study is to determine if a Contura catheter can avoid a radiation "hot spot" in the skin and improve tissue-balloon conformance in early-stage breast cancer patients undergoing accelerated partial breast irradiation.

DETAILED DESCRIPTION:
In approximately 20% of patients who are considered for accelerated partial breast irradiation (APBI), the balloon-to-skin distance ranges from 3-6 mm. The Contura applicator has 5 source lumens. In contrast, the MammoSite catheter has a single source lumen. The ability to choose from multiple source lumens with the Contura catheter allows one to avoid a radiation "hot spot" in the skin in cases where the balloon-to-skin spacing is only 3-6 mm.

Another limitation of the MammoSite catheter is that one cannot improve on the suboptimal conformance of the balloon with the surrounding breast tissue. An air/fluid pocket next to the balloon can push breast tissue at greatest risk of harboring residual disease away from the radioactive source. With APBI, the planning target volume for plan evaluation (PTV_EVAL) is defined as the breast tissue volume bounded by uniform expansion of the balloon radius in all dimensions by 10 mm less the balloon volume. PTV_EVAL is limited to 5 mm from the skin surface and by the posterior breast tissue extent (chest wall and pectoralis muscles are excluded). The volume of an air/fluid pocket is usually 4.8% ± 1.1% (mean ± standard error) of PTV_EVAL. The Contura applicator has a vacuum lumen with 2 openings adjacent to the balloon that allow for air/fluid removal. By using the vacuum lumen on a Contura applicator, one can typically decrease the size of an air/fluid pocket by about one third. In approximately 90% of Contura patients, the volume of an air/fluid pocket around the balloon can be reduced to less than or equal to 3.0% of PTV_EVAL. In contrast, the volume of an air/fluid pocket around the balloon is less than or equal to 3.0% of PTV_EVAL in only about half of MammoSite patients. Since this study addresses intermediate-risk patients, it is particularly important that the size of an air/fluid pocket be minimized with a Contura applicator.

SenoRx, Inc. (Aliso Viejo, CA) is currently conducting a registry study of the Contura MLB applicator in the "low-risk" patient population. This "intermediate-risk" study is complimentary to the low-risk registry study. There is no overlap in patient eligibility. Intermediate-risk patients meet any of the following criteria:

1. Age 18-49 years, or
2. Estrogen receptor-negative and progesterone receptor-negative breast cancer, or
3. 1-3 involved axillary lymph nodes

ELIGIBILITY:
Inclusion Criteria:

* Patients with invasive breast cancer are required to have axillary staging which can include sentinel node biopsy alone if sentinel node is negative or axillary dissection or sampling with a minimum total of 6 axillary nodes if sentinel node is positive. Axillary staging is not required for patients with DCIS.
* Estrogen receptor (ER) and progesterone receptor (PR) analysis must be negative.
* The patient must be ≥ 18 years old.
* If the patient is older than 49 years, she must meet at least one of the following 2 conditions:

  i. 1-3 histologically positive axillary nodes ii. negative ER and PR analysis
* The patient should have a life expectancy of at least 10 years, excluding her diagnosis of breast cancer.
* The tumor must be DCIS or invasive adenocarcinoma of the breast.
* Gross disease must be unifocal with pathologic tumor size 3.0 cm or less. Patients with microscopic multifocality are eligible as long as total pathologic tumor size is 3.0 cm or less.
* The patient must have pathological stage 0, I, or II breast cancer.
* Surgical treatment of the breast must have been lumpectomy. The margins of the resected specimen must be histologically free of tumor (DCIS and invasive). Re-excision of surgical margins is permitted.
* The patient must be registered within 42 days following the last surgery for breast cancer.
* The target lumpectomy cavity/whole breast reference volume must be ≤ 30% based on the postoperative CT scan.

Exclusion Criteria:

* The patient is < 18 years old.
* If the patient is older than 49 years, she has both an ER and PR positive tumor and histologically negative axillary nodes.
* T2 (> 3.0 cm), T3, stage III, or stage IV breast cancer.
* "Marginal" or "borderline" ER or PR analysis results.
* More than 3 histologically positive axillary nodes.
* Axillary nodes with definite evidence of microscopic or macroscopic extracapsular extension.
* One or more positive non-axillary sentinel node(s). Intramammary nodes are staged as axillary nodes.
* Non-epithelial breast malignancies such as sarcoma or lymphoma.
* Proven multicentric carcinoma in more than one quadrant or separated by 4 or more centimeters.
* Paget's disease of the nipple.
* Synchronous bilateral invasive or non-invasive breast cancer.
* History of DCIS or invasive breast cancer.
* Surgical margins that cannot be microscopically assessed or are positive at pathologic evaluation.
* Clear delineation of the target lumpectomy cavity not possible.
* Any treatment with radiation therapy, chemotherapy, and/or biotherapy administered for the currently diagnosed breast cancer prior to registration. The only exception is hormonal therapy, which may have been given for no more than a total of 28 days anytime after diagnosis and before registration.
* Prior breast or thoracic radiotherapy for any condition.
* Collagen vascular disease, specifically dermatomyositis with a CPK level above normal or with an active skin rash, systemic lupus erythematosis, or scleroderma.
* Pregnancy or lactation at the time of proposed registration. Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy.
* Psychiatric or addictive disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Maximum skin dose is less than or equal to 100% of the prescribed radiation dose and air/fluid pocket next to the balloon is less than or equal to 3.0% of the planning target volume for plan evaluation | 19 months

SECONDARY OUTCOMES:
Number of cases where the balloon catheter has to be explanted when the balloon-to-skin spacing is only 3-6 mm. | 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Wilder, MD, Principal Investigator — Cancer Center of Irvine; Kenneth M Tokita, MD, Study Chair — Cancer Center of Irvine
Locations (1):
- Cancer Center of Irvine, Irvine, California, United States